CLINICAL TRIAL: NCT02004717
Title: Phase 1, Open-label Study to Assess the Safety, Tolerability, and Pharmacokinetics of DS-8895a in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Study of DS-8895a in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8895-A-J101
Record Dates: First submitted 2013-11-15; First posted 2013-12-09 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumors
Keywords: advanced solid tumor; Phase 1; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose escalation then expansion (Experimental): Dose escalation of this study will follow a 3+3 study design with a starting intravenous (IV) dose of 0.1 mg/kg. Six dose levels are planned: level 1,0.1 mg/kg; level 2,0.3 mg/kg; level 3, 1.0 mg/kg; level 4,3.0 mg/kg; level 5,10 mg/kg; level 6,20 mg/kg.
  Dose Expansion - Up to 20 subjects will be enrolled and treated at the dose determined in Dose Escalation arm.
  Interventions: Drug: DS-8895a

INTERVENTIONS:
Drug: DS-8895a

SUMMARY:
This is an open-label, sequential dose escalation and expansion study to evaluate the safety, tolerability, and pharmacokinetics of DS-8895a in Japanese subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor that is refractory to standard treatment, or for which no standard treatment is available.
* Eastern Cooperative Oncology Group performance status(PS) of 0 or 1

Exclusion Criteria:

* Have any of the following concomitant disease or had the history of having following disease within 6 months before enrollment:

Cardiac failure (NYHA ≥ ClassIII), myocardial infarction, cerebral infarction, unstable angina, arrhythmia requiring treatment, coronary-artery/peripheral artery bypass surgery, cerebrovascular disease, pulmonary thromboembolism, deep-vein thrombosis or clinically severe thromboembolic event, or clinically severe pulmonary disease (eg, interstitial pneumonia, pulmonary fibrosis, radiation pneumonia, drug induced pneumonia)

* Severe or uncontrolled concomitant disease.
* Clinically active brain metastases defined as symptomatic or requiring treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
number of participants experiencing dose limiting toxicities | day 1 through day 28
  to investigate the safety of DS-8895a reporting on frequency and seriousness of treatment emergent adverse events
number of participants experiencing clinical or laboratory adverse events | from start of treatment to end of treatment, on expected average 12 weeks
  to investigate the safety of DS-8895a reporting on frequency and seriousness of treatment emergent adverse events
serum pharmacokinetics of DS-8895a | Cycle 1 - days 1, 2, 4, 8 and 15; Cycle 2-days 1, 2, 4, 8 and 15; Cycle 3 and on- days 1; end of study; 45 days post last dose
  pharmacokinetics (Area Under the Curve-AUC, Terminal Elimination half-life-t1/2, Total Body Clearance) of DS-8895a in Japanese subjects with advanced solid tumors, and also to investigate the recommended dose of DS-8895a for subsequent clinical studies

SECONDARY OUTCOMES:
level of anti-DS-8895a (HAHA) antibody | Cycle 1 days 1 and 15; Cycle 2 day 1; end of study; 45 days post-last-dose
  Human anti-human antibody (HAHA) profile for DS-8895a [Time Frame: Cycle 1 - days 1, and 15; Cycle 2 and on - days 1; end of study; 45 days post last dose] The presence of HAHA (anti-DS-8895a neutralizing antibody) in serum will be assessed"
disease control rate | every 6 weeks
  proportion of subjects with the best overall response of stable disease or better will be measured every 6 weeks until study drug discontinued.
pharmacodynamic effects in blood | day 1 and 2
  effects on blood will be determined at day 1 and 2 of each cycle
pharmacodynamic effects in tumors | baseline and day 1 of cycle 2
  effects on tumor cells will be determined at baseline and day 1 of cycle 2
objective response rate | every 6 weeks
  sum of complete response and partial response rates measured every 6 weeks until study drug discontinuation

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Osaka University Hospital, Suita, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shitara K, Satoh T, Iwasa S, Yamaguchi K, Muro K, Komatsu Y, Nishina T, Esaki T, Hasegawa J, Kakurai Y, Kamiyama E, Nakata T, Nakamura K, Sakaki H, Hyodo I. Safety, tolerability, pharmacokinetics, and pharmacodynamics of the afucosylated, humanized anti-EPHA2 antibody DS-8895a: a first-in-human phase I dose escalation and dose expansion study in patients with advanced solid tumors. J Immunother Cancer. 2019 Aug 14;7(1):219. doi: 10.1186/s40425-019-0679-9. PMID 31412935